CLINICAL TRIAL: NCT03624231
Title: Ph II Trial to Assess Feasibility+Efficacy of Treatment w Durva+Treme+Radiation and Treatment w Durva+Radiation as First-line Therapy for Patients w Non-resectable Locally Advanced HPV-HNSCC- a Comparision With a Historical Control Group
Brief Title: Feasibility & Efficacy of Durvalumab+Tremelimumab+RT and Durvalumab+RT in Non-resect. Locally Advanced HPVnegativ HNSCC
Acronym: DURTRE-RAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ulrich Keilholz (Other)
Collaborators: Charite University, Berlin, Germany (Other); AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Ulrich Keilholz, Director of the Charité Comprehensive Cancer Center, Principal Investigator, Clinical Professor, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DURTRE-RAD
Record Dates: First submitted 2017-12-05; First posted 2018-08-10 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — durvalumab; tremelimumab; Radiotherapy

STUDY DESIGN:
Intervention Model Description: 2-arm, randomized, multicenter, phase II. Step 1 is Registration. All patients need to sign the informed consent form for registration. Tumor tissue then be send to the central lab for defining the HPV status. If the patient is HPV negative the site will be notified if they can further proceed to patient randomization.
  Step 2 is Randomization of all eligible patients with a centrally diagnosed, HPV negative tumor one of the two arms Durvalumab plus Tremelimumab + radiotherapy; Durvalumab + radiotherapy) after signing the informed consent form for step 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - stopped after interims analyses (Experimental): Patients in arm 1 will receive a single dose of durvalumab of 1500 mg administered on day 1, 14 days prior to initiation of the radiotherapy.
  Radiotherapy with 35 fractions over 7 weeks (administered as daily fractions of 2 Gy given 5 days every week for 7 weeks) will start on day 14. On week 5, 9, 13 and 17 patients will receive durvalumab (1500 mg) and tremelimumab (75 mg) for up to 4 doses/cycles and then continue 1500 mg durvalumab q4w starting on week 21 to complete a total of 12 months of therapy (overall 9 single doses durvalumab including the initial dose on day 1).
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Radiation: Radiotherapy
- Arm 2 (Experimental): Patients in arm 2 will receive durvalumab (1500 mg) q4w starting on day 1. Radiotherapy with 35 fractions over 7 weeks (administered as daily fractions of 2 Gy given 5 days every week for 7 weeks) will start on day 14.
  Overall patients will receive treatment with durvalumab mono up to a total of 12 months (up to 13 doses in total).
  Interventions: Drug: Durvalumab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Durvalumab — Durvalumab (1500 mg) starting on week 1 to complete a total of 12 months
  Other Names: MEDI4736
Drug: Tremelimumab — Tremelimumab (75 mg) for up to 4 doses/cycles
  Arms: Arm 1 - stopped after interims analyses
Radiation: Radiotherapy — Radiotherapy with 35 fractions (administered as daily fractions of 2 Gy given 5 days every week for 7 weeks)

SUMMARY:
Phase II trial evaluating to assess the feasibility and efficacy as first-line therapy for patients with non-resectable locally advanced HPV negative HNSCC of Durvalumab a PDL1-Inhibitor plus Tremelimumab a CTLA-4- Inhibitor in combination with radiotherapy and Durvalumab in combination with radiotherapy as first-line therapy.

2-arm, randomized, multicenter, phase II. Step 1 is Registration. All patients need to sign the informed consent form for registration. Tumor tissue then be send to the central lab for defining the HPV status. If the patient is HPV negative the site will be notified if they can further proceed to patient randomization.

Step 2 is Randomization of all eligible patients with a centrally diagnosed, HPV negative tumor in one of the two arms (Durvalumab plus Tremelimumab + radiotherapy; Durvalumab + radiotherapy) after signing the informed consent form for step 2.

DETAILED DESCRIPTION:
The primary objective is to explore the feasibility and efficacy in terms of treatment discontinuation due to toxicity and in terms of 1-year progression free survival of a PDL1-Inhibitor plus a CTLA-4 Inhibitor in combination with radiotherapy and a PDL1-Inhibitor in combination with radiotherapy as first-line therapy for patients with non-resectable locally advanced HNSCC in the poor prognostic subgroup.

Secondary objectives are to investigate the benefit of the addition of a CTLA-4 Inhibitor and/or a PDL1-Inhibitor to radiotherapy in terms of overall progression free survival, overall survival and to investigate the approach in terms of safety, chronic toxicity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced histopathologically confirmed HNSCC not candidate for primary surgical treatment
* No distant metastasis (M0)
* Tumor tissue available for central testing Patient with HPV/p16 negative disease (≤70% positively stained cells) as determined by central testing
* Adequate normal organ and marrow function
* Measurable tumor according to RECIST
* Patients must be expected to complete the treatment.
* Age > 18 years at time of study entry
* Female patients must either be of non-reproductive potential or must have a negative serum pregnancy test upon study entry and be willing to use adequate contraceptive measurements as described in the protocol
* Non-sterilized males who are sexually active with a female partner of childbearing potential must be willing to use adequate contraceptive measurements as described in the protocol section 6.5.4

Exclusion Criteria:

* Participation in another clinical study with an investigational product during the last 3 months
* Prior or current anticancer treatment to the head and neck area (e.g. radical attempted or tumor reductive surgery, neo-adjuvant chemotherapy, EGFR inhibitors or radiotherapy).
* Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab or an anti-CTLA4, including tremelimumab
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone History of primary immunodeficiency
* History of allogeneic organ transplant
* History of another primary malignancy except for

  * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* History of hypersensitivity to durvalumab and/or tremelimumab or any excipient
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control as described in the protocol from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period
* Distant metastasis
* Patients who are institutionalised by official order
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fredericia's Correction
* Receipt of live attenuated vaccination within 30 days prior to study entry step 2 or within 30 days of receiving durvalumab or tremelimumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Efficacy- 1-year progression free survival (PFS) | 1 year
  1-year progression free survival (PFS) depicted as the 1-year in-field-progression-free survival and 1-year distant metastasis free survival
Feasibility - Number of treatment discontinuations due to toxicity | During treatment
  number of treatment discontinuations due to toxicity

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of randomization until the date of death, assessed up to 3 years
  defined as the time from patient inclusion to the date of death or date of last follow-up news
Safety - Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | From date of randomization until the date of study assessed up to 3 years
  defined as event possibly related to study treatment and fulfills the criteria using CTCAE Version 4.03
Chronic toxicity -Number of participants with treatment-related adverse Events Lasting longer than 3 months as assessed by CTCAE v4.03 and/or RTOG/EORTC Late Radiation Morbidity Scoring Schema | From date of randomization until the date of study assessed up to 3 years
  defined as event lasting longer than 3 months and possibly related to study treatment and fulfills the criteria using CTCAE Version 4.03 and/or and/or RTOG/EORTC Late Radiation Morbidity Scoring Schema
Quality of life (QoL) - measured by EORTC QLQ-H&N35 and EORTC QLQ-C30) | From date of randomization until the date of study assessed up to 3 years
  defined as assessment for evaluation of medical and psychosocial interventions

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Keilholz, MD, Study Chair — Charité Comprehensive Cancer Center
Locations (3):
- Germany (3):
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Vivantes Klinikum Neukölln, Berlin
  - Charité Comprehensive Cancer Center, Berlin

IPD SHARING:
Plan to Share IPD: No